CLINICAL TRIAL: NCT02336152
Title: Use of Onepiece Suit or Forced Warm Air for Perioperative Temperature Conservation.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Varmedrakt.OUS.15.1
Record Dates: First submitted 2015-01-05; First posted 2015-01-12 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Surgery
MeSH Terms: interventions — Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Body suit (Experimental): The patients will receive a body suit at least 30 min before start of general anaesthesia, and will keep the suit on until warm and comfortable in the post-operative unit. The suit is supplied with multiple snap openings to allow for draping, washing and surgery.
  Interventions: Device: Anaesthesia, Teles Pro, Body suit
- Forced warm air (Active Comparator): The patients will receive forced warm air on their lower body when placed on operating table, ready for surgery.
  Interventions: Device: Anaesthesia, Teles Pro, Body suit

INTERVENTIONS:
Device: Anaesthesia, Teles Pro, Body suit

SUMMARY:
To study if a one piece body suite (T-balance, Telespro, Finland) is equally effective in maintaining peri-operative body temperature as forced air warming, during open low-back surgery of medium duration.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3
* Approved consent
* Expected duration of open back surgery of 60-120 min
* Prestudy core temperature (oral) of at least 36 degrees C

Exclusion Criteria:

* Known diabetes mellitus
* Any known illness or use of pre-op drugs which may interfere with normal temperature regulation
* Body mass index less than 17 or more than 35
* Pregnancy
* Any contraindication for warming device or temperature monitor

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-06 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Body core temperature | 30 minutes after anaesthesia induction
  SpotOn (3M) measurement in the forehead

SECONDARY OUTCOMES:
Body core temperature | 1 hr before - intraoperative - 3 hrs postoperative
Patient termal satisfaction | 1 hr before - intraoperative - 3 hrs postoperative
  patient interview

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Anesthesiology, Oslo University Hospital, Ullevaal, Oslo, Norway